CLINICAL TRIAL: NCT04504370
Title: A Phase III, Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Pegylated Exenatine Injection (PB-119) in Drug-naïve T2DM Subjects
Brief Title: Safety and Efficacy of Pegylated Exenatine Injection (PB-119) in Drug-naïve T2DM Subjects
Acronym: PB119
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB119301
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-119 once-weekly-subcutaneous injection (Experimental): PB119 (polyethylene glycol exenatide) is a long-acting GLP-1RA for injection, which will be administered 150μg once-weekly subcutaneously to patients in active drug group for 24 weeks.
  Interventions: Drug: GLP-1 receptor agonist
- Placebo once-weekly-subcutaneous injection (Placebo Comparator): PB-119 150μg matched placebo which will be used in placebo group for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-1 receptor agonist — PB-119 is an investigational pegylated human glucagon-like peptide-1 (GLP-1) receptor agonist. The dosing regimen is 150μg once every week as subcutaneous administration. Patients in PB-119 group will be administered the active drugs for 52 weeks (24+28).
  Arms: PB-119 once-weekly-subcutaneous injection
Drug: Placebo — PB-119 matched placebo will be used once every week as subcutaneous administration to placebo group for 24 weeks.
  Other Names: PB-119 Placebo
  Arms: Placebo once-weekly-subcutaneous injection

SUMMARY:
A randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of 24 once-weekly subcutaneous doses of PB-119 in Drug-naïve T2DM Subjects.

DETAILED DESCRIPTION:
The study included a maximum 2-week screening period, a 4-week single-blind introduction period, a 24-week double-blind treatment period, a 28-week open extension treatment period, and a 4-week safety follow-up period.

At the end of the single-blind entry period, eligible subjects were randomly assigned to two different administration groups in a 1:1 ratio and received a 24-week double-blind treatment.

All subjects who completed the double-blind treatment entered the open extension treatment phase.Open extension treatment with subcutaneous injection of 150μg PB-119 once a week for 28 weeks.

Safety follow-up was conducted 4 weeks after the end of treatment/completion of early exit visit in the open extension period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18~75 years old;
* Confirmed T2DM patients meet the diagnostic criteria for type 2 diabetes published by WHO1999；
* 18.5 kg/m2 < BMI < 40.0 kg/m2 at screening;
* 7.5% ≤ HbA1c ≤ 11.0% at screening;
* 7.0% ≤ HbA1c ≤ 10.5% when the random;
* 18.5 kg/m2 < BMI < 40.0 kg/m2 during screening and before randomization

Exclusion Criteria:

* T1DM;
* Continuous use of insulin for more than 14 days within 1 year before screening or before randomization；
* Treatment with any dipeptidylpeptidase 4 (DPP-4) inhibitor or glucose-dependent insulin-stimulating peptide (GIP) or/and glucagon-like peptide-1 (GLP-1) receptor agonist prior to screening or randomized prior treatment；
* Screening for any of the following heart diseases within the first 6 months or before randomization；
* Patients whose hypertension was not effectively controlled during screening or before randomization (after resting ≥5 minutes, systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg)；
* Serum amylase or lipase >3×ULN or those with previous diagnosis of acute/chronic pancreatitis were screened or randomly screened；
* Screening for severe trauma or infection that may affect glycemic control within the first month or before randomization；
* A history or family history of medullary thyroid carcinoma (MTC) or multiple endocrine adenomatosis type 2 (MEN2)；
* Known to be allergic or intolerant to the study drug or metformin；
* Female subjects during pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | week 1, week 25
  Change in HbA1c from baseline(week 1) to week 25

SECONDARY OUTCOMES:
HbA1c Below 7.0% | week 1, week 25
  Percentage of participants with HbA1c below 7.0% was evaluated at week 25.
Change in Body Weight (kg) | week 1, week 25
  Change from baseline (week 1) in body weight was evaluated at week 25
Change in Fasting Plasma Glucose (FPG) | week 1, week 25
  Change from baseline (week 1) in FPG was evaluated at week 25
Change in Body Mass Index | week 1, week 25
  Change from baseline (week 1) in body mass index (BMI) was evaluated at week 25.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD,PhD, Principal Investigator — Central South University The Second Xiangya Hospital; WeiHong Song, MD,PhD, Principal Investigator — First People's Hospital of Chenzhou; Jing Yang, MD,PhD, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Bin Gao, MD,PhD, Principal Investigator — Tang-Du Hospital; Lin Liao, MD,PhD, Principal Investigator — Qianfoshan Hospital; YanJun Wang, MD,PhD, Principal Investigator — Second Hospital of Jilin University; Minxiu Yao, MD,PhD, Principal Investigator — Qingdao Central Hospital; Huige Shao, MD,PhD, Principal Investigator — Changsha Central Hospital; Jingna Lin, MD,PhD, Principal Investigator — Tianjin People's Hospital; Jiarui Li, MD,PhD, Principal Investigator — Cangzhou Central Hospital; Xiaohong Lin, MD,PhD, Principal Investigator — ZhuZhou Central Hospital; Guixia Wang, MD,PhD, Principal Investigator — The First Hospital of Jilin University; Jianhua Ma, MD,PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Zhinong Zhang, MD,PhD, Principal Investigator — Qiqihar First Hospital
Locations (1):
- Central South University The Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan X, Ma J, Liu Y, Wang X, Li S, Yan S, Mo Z, Zhu Y, Lin J, Liu J, Jia Y, Liu L, Ding K, Xu M, Zhou Z. Efficacy and safety of visepegenatide, a long-acting weekly GLP-1 receptor agonist as monotherapy in type 2 diabetes mellitus: a randomised, double-blind, parallel, placebo-controlled phase 3 trial. Lancet Reg Health West Pac. 2024 Jun 7;47:101101. doi: 10.1016/j.lanwpc.2024.101101. eCollection 2024 Jun. PMID 38948164